CLINICAL TRIAL: NCT01242332
Title: Perioperative Administration of Pregabalin in Patients Undergoing Arthroscopic Anterior Cruciate Ligament Reconstruction: Does it Help to Relieve Postoperative Pain?
Brief Title: Perioperative Administration of Pregabalin in Patients Undergoing Arthroscopic Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Sasikaan Nimmaanrat, Dr. (MD), Deparment of Anesthesiology, Faculty of Medicine, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC 52 -234-08-1-2
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2009-05

CONDITIONS: Postoperative Pain Management
Keywords: perioperative; pregabalin; arthroscopic anterior cruciate ligament reconstruction; postoperative pain management
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (No Intervention): po 2 hrs before surgery
- Pregabalin (Experimental): 75 mg po 2 hrs before surgery
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — 75 mg po 2 hrs before surgery
  Other Names: Lyrica
  Arms: Pregabalin

SUMMARY:
To prove pregabalin's efficacy and safety in Thai patients scheduled for arthroscopic ACL reconstruction

DETAILED DESCRIPTION:
Only eligible patients with willingness to join this study are included. Eligible patients are those aged 18-65 years of either sex, American Society of Anesthesiologists (ASA) physical status I & II, and body mass index (BMI) between 16-35. The exclusion criteria are patients who are allergic to pregabalin, with impaired hepatic and renal functions, alcohol or substance abuse, chronic pain (except pain in the knee joint) or daily intake of analgesics, uncontrolled medical disease (hypertension and diabetes mellitus) and inability to operate patient-controlled analgesia (PCA) device.

Data analysis

* Student t-test for continuous data with normal distribution
* Mann-Whitney U test for continuous data with non-normal distribution
* Chi-square test for categorical data

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are those aged 18-65 years of either sex,
* American Society of Anesthesiologists (ASA) physical status I & II, and body mass index (BMI) between 16-35.

Exclusion Criteria:

* patients who are allergic to pregabalin,
* impaired hepatic and renal functions,
* alcohol or substance abuse,
* chronic pain (except pain in the knee joint) or daily intake of analgesics, uncontrolled medical disease (hypertension and diabetes mellitus)
* inability to operate patient-controlled analgesia (PCA) device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
efficacy | August 2009 - January 2011
  efficacy of postoperative pain management

SECONDARY OUTCOMES:
safety | August 2009 - January 2011
  safety of pregabalin for postoperative pain management

CONTACTS AND LOCATIONS:
Overall Officials: Sasikaan Nimmaanrat, MD, MMed, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Prince of Songkla University
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

REFERENCES:
- [Result] Chang SH, Lee HW, Kim HK, Kim SH, Kim DK. An evaluation of perioperative pregabalin for prevention and attenuation of postoperative shoulder pain after laparoscopic cholecystectomy. Anesth Analg. 2009 Oct;109(4):1284-6. doi: 10.1213/ane.0b013e3181b4874d. Epub 2009 Jul 29. PMID 19641054